CLINICAL TRIAL: NCT06772844
Title: DNA Methylation Analysis in Stool Samples for Screening of Lynch Syndrome-Associated Colorectal Cancer
Brief Title: DYNAMICS-LYNCH：DNA Methylation Analysis in Stool for Screening of Lynch Syndrome-Associated Colorectal Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Pei-Rong Ding, director, Sun Yat-sen University
Other Study IDs: 2024-FXY-142
Record Dates: First submitted 2025-01-10; First posted 2025-01-14 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Colorectal Cancer Screening; Lynch Syndrome
Keywords: lynch syndrome; colorectal cancer; screening
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — stool
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with lynch syndrome: Patients diagnosed with Lynch syndrome by genetic testing
  Interventions: Diagnostic Test: fecal DNA methylation testing

INTERVENTIONS:
Diagnostic Test: fecal DNA methylation testing — Three rounds of screening were performed. In the first year, colonoscopy was conducted along with concurrent fecal DNA testing performed prior to the colonoscopy. In the second year, fecal DNA testing was performed only if no polyps were detected during the colonoscopy in the first year; otherwise, both colonoscopy and fecal DNA testing were conducted. In the third year, a colonoscopy was performed with concurrent fecal DNA testing conducted before the procedure

SUMMARY:
Colorectal cancer (CRC) has high incidence and mortality rates globally. Over 1 million new cases are diagnosed annually, and about 600,000 people die from the disease each year. In China, CRC ranks third in incidence and fifth in mortality. Its rates are rising due to lifestyle changes and an aging population.

Around 30% of CRC cases have a hereditary component, including familial adenomatous polyposis (FAP) and Lynch syndrome. Lynch syndrome, or hereditary non-polyposis colorectal cancer (HNPCC), accounts for 3%-5% of CRC cases. Early diagnosis, screening, and prophylactic surgery can reduce CRC mortality by 7%-42%, and mortality from endometrial and ovarian cancers by 1%-6%. Intensive screening is essential for Lynch syndrome patients, who are at high risk for CRC.

Due to the lack of early symptoms, many CRC cases are diagnosed in later stages, causing financial strain on patients, families, and society. Screening is an effective tool in reducing CRC-related mortality by more than 50%. In developed countries such as the U.S., U.K., and Japan, CRC screening is integrated into public health programs, emphasizing its role in prevention.

In China, CRC screening mainly involves the fecal occult blood test followed by colonoscopy, but this method faces challenges. First, the fecal occult blood test lacks sufficient sensitivity, leading to underdiagnosis. Second, colonoscopy is invasive with low patient acceptance. It also requires specialized facilities, advanced equipment, and skilled endoscopists, limiting its accessibility. Given China's large population and limited healthcare resources, universal colonoscopy screening is challenging, resulting in low screening rates.

To address these challenges, we propose replacing part of colonoscopy screening with DNA methylation testing of fecal samples. Self-sampling methylation screening could ease the strain on healthcare resources and improve patient compliance. By combining methylation screening with colonoscopy, we aim to reduce colonoscopy frequency and enhance overall compliance.

This study will include three rounds of methylation screening with colonoscopy as the control, involving 400 Lynch syndrome patients. The goal is to develop new screening criteria for this high-risk group, reduce colonoscopy frequency, and ultimately lower CRC incidence in Lynch syndrome patients.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is a malignant disease with a high incidence and mortality rate worldwide. Globally, more than 1 million new cases of CRC are diagnosed annually, and approximately 600,000 patients die from the disease each year. In China, CRC has the third-highest incidence, following lung and stomach cancers and the fifth-highest mortality rate. With changes in lifestyle and an aging population, the incidence and mortality rates of CRC in China have been continuously rising. About 30% of colorectal cancer (CRC) patients exhibit a hereditary predisposition, including familial adenomatous polyposis (FAP) and Lynch syndrome. Lynch syndrome, also known as hereditary non-polyposis colorectal cancer (HNPCC), is the most common hereditary colorectal cancer, accounting for 3%-5% of CRC cases. Several clinical criteria, such as the Amsterdam Criteria and Bethesda guidelines, are applied to the diagnosis of Lynch syndrome. Effective diagnosis, screening, and prophylactic surgery for Lynch syndrome can significantly reduce colorectal cancer mortality by 7%-42%, as well as mortality from endometrial and ovarian cancers by 1%-6%. Intensive screening measures are critical for patients with Lynch syndrome, who are considered to be at high-risk for CRC.

Due to the lack of early symptoms, many CRC patients are diagnosed at the middle to late stages of the disease, which places significant financial pressure not only on the patients themselves but also on society and their families. Screening is one of the most effective tools for preventing colorectal cancer and can reduce mortality by more than 50%. In developed countries such as the United States, the United Kingdom, and Japan, colorectal cancer screening has been integrated into public health programs, highlighting its critical role in disease prevention. Currently, colorectal cancer screening relies on the fecal occult blood test, followed by detailed examinations such as colonoscopy in our country, which still presents several challenges. First, the sensitivity of the fecal occult blood test is insufficient, leading to a high rate of underdiagnosis. Second, colonoscopy is an invasive procedure with relatively low acceptance among patients. Furthermore, colonoscopy is typically performed in a facility-based setting, which requires advanced endoscopic equipment and experienced endoscopists, making it highly dependent on medical resources. Given the limited healthcare resources, achieving universal coverage of the entire population with a facility-centered colonoscopy model is challenging, resulting in a low overall screening rate. Improvements are needed to enhance the efficiency and coverage of screening programs to better prevent and control the incidence of CRC. For patients with Lynch syndrome, intensive colonoscopy may lead to poor compliance due to its tedious process. To address these challenges, we propose to replace part of the colonoscopy screening with DNA methylation testing for fecal samples. Self-sampling methylation screening for colorectal cancer in patients with Lynch syndrome could not only alleviate the excessive strain on healthcare resources but also improve patient compliance with screening.

To explore the optimal screening strategy, reduce the frequency of colonoscopy, and improve patient compliance, we propose conducting methylation screening alongside colonoscopy for patients with Lynch syndrome. This study will include three consecutive rounds of head-to-head methylation screening, with colonoscopy as the control, involving 400 patients with Lynch syndrome. We aim to identify new screening criteria for this high-risk group, reduce the frequency of colonoscopy, improve screening compliance, and ultimately reduce the incidence of colorectal cancer in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent: patients are required to participate voluntarily and sign an informed consent form in writing；Patients diagnosed with Lynch syndrome；Agree to collect and send stool specimens for methylation sequencing as required；Willingness to undergo long-term follow-up and three rounds of methylation screening

Exclusion Criteria:

* Patients with confirmed familial adenomatous polyposis or other hereditary colorectal cancers that are not Lynch syndrome；Patients who are unable to obtain a fecal specimen or whose specimen is substandard for follow-up testing；Patients diagnosed with colorectal cancer or currently undergoing surgery；Failure to sign informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients attending Sun Yat-sen University Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-01-10 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Receiver Operating Characteristic Curve | From enrollment to the end of test at 3years
  Area Under the Curve（AUC）